CLINICAL TRIAL: NCT03803579
Title: Baseline DOAC Measurement in Non Valvular Atrial Fibrillation Patients and Incidence of Bleeding or Thromboembolic Complications During Follow-up: a Prospective, Multicenter, Observational Study. The MAS (Measure And See) Study
Brief Title: Baseline Concentration of Direct Oral Anticoagulant and Incidence of Adverse Event Measure And See (MAS)
Acronym: MAS
Status: Completed | Type: Observational
Sponsor: Arianna Anticoagulazione Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: FAA O3 12-2017 (MAS)
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation; Anticoagulant-induced Bleeding
Keywords: Atrial Fibrillation; Bleeding event; Thromboembolic event; Plasma concentration of drug
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MAS Study is an observational, multicentre, prospective cohort study in Non valvular Atrial fibrillation (NVAF) patients treated with one of the direct oral anticoagulants (DOACs) available in Italy for NVAF patients.

The general aim is to deepen the knowledge of DOAC treatment in NVAF patients, by measuring the plasma concentration of anticoagulant drugs and their correlation with any adverse events that may occur during treatment.

DETAILED DESCRIPTION:
The MAS Study is an observational, prospective cohort study, double blind, multicentre, international and no Profit. Anticoagulation clinics, affiliated or not to the Italian FCSA, will be asked to take an active part in the study, provided they have the facilities for blood sampling and processing.

4000 consecutive NVAF outpatients, 1000 for each single drug, starting anticoagulation with one of the four DOAC (apixaban, dabigatran, edoxaban, rivaroxaban) will be enrolled at the moment of the first prescription. Patients will receive the type and dosage of DOAC on the base of clinical characteristics at the discretion of the attending physician, as the normal clinical practice, and the study will not influence the decision of the type and dosage of DOAC.

The primary study objective is to evaluate the possible relationship between DOAC anticoagulant levels at the trough, measured at steady state (within the first 2-4 weeks of treatment) and occurrence of bleeding and thromboembolic events during the subsequent one year follow up

ELIGIBILITY:
Inclusion Criteria:

* NVAF patients starting DOAC anticoagulation
* age > 18 years
* ability to give written informed consent
* availability, as part of the normal withdrawals, to the blood sampling for the study purpose
* availability for 12-months follow-up

Exclusion Criteria:

* age < 18 years
* indication for electrical cardioversion at the moment of drug prescription
* participation in Phase II or III clinical trials
* indication for treatment different from NVAF
* not suitable to give or not giving informed consent
* not available for blood collection or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4000 consecutive Non Valvular Atrial Fibrillation outpatients, 1000 for each single drug, aged >18 years and starting anticoagulation with one of the four DOAC (apixaban, dabigatran, edoxaban, rivaroxaban) will be enrolled at the moment of the first prescription. Patients will receive the type and dosage of DOAC on the base of clinical characteristics at the discretion of the attending physician, as the normal clinical practice, and the study will not influence the decision of the type and dosage of DOAC
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Number and rate of major bleeding events and clinically relevant bleeds (defined according to International Society on Thrombosis and Haemostasis guidelines) | From date of enrollment until the date of first documented event assessed up to 12 months
  Fatal bleeding; Acute clinically overt bleeding;intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal will be recorded in all patients.
Number and rate of patients with confirmed thromboembolic and thromboembolic-related dath | From date of enrollment until the date of first documented event assessed up to 12 months
  Cardiovascular event: transient ischemic attack, stroke. myocardial infarction; the occurrence of deep vein thrombosis with or without pulmonary embolism will be recorded in all patients.
Number and rate of death patients (overall mortality) | From date of enrollment until the date of first documented event assessed up to 12 months
  Cardiovascular related death; thromboembolic related dath, bleeding-related death, cancer related death will be recorded in all patients
Through plasma concentration (ng/ml) of Apixaban, Dabigatran, Edoxaban and Rivaroxaban | 15-20 days after the enrollment
  Blood sampling is performed at trough level for each anticoagulant drug used after the last dose intake of dabigatran, apixaban, rivaroxaban and edoxaban

SECONDARY OUTCOMES:
Number and rate of patients who discontinued treatment | From date of enrollment until the date of first documented event assessed up to 12 months
  The treatment withdrawal, either for patients or for physician decision-making will be recorded in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Testa, MD, Study Director — UUOO Lab Analisi Chim Cliniche Microb-Centro Emostasi, ASST-Cremona Italy
Locations (1):
- Sophie Testa, Cremona, Italy

REFERENCES:
- [Derived] Palareti G, Testa S, Legnani C, Dellanoce C, Cini M, Paoletti O, Ciampa A, Antonucci E, Poli D, Morandini R, Tala M, Chiarugi P, Santoro RC, Iannone AM, De Candia E, Pignatelli P, Faioni EM, Chistolini A, Esteban MDP, Marietta M, Tripodi A, Tosetto A. More early bleeds associated with high baseline direct oral anticoagulant levels in atrial fibrillation: the MAS study. Blood Adv. 2024 Sep 24;8(18):4913-4923. doi: 10.1182/bloodadvances.2024013126. PMID 38842448
- [Derived] Testa S, Palareti G, Legnani C, Dellanoce C, Cini M, Paoletti O, Ciampa A, Antonucci E, Poli D, Morandini R, Tala M, Chiarugi P, Santoro RC, Iannone AM, De Candia E, Pignatelli P, Faioni EM, Chistolini A, Esteban MDP, Marietta M, Tripodi A, Tosetto A. Thrombotic events associated with low baseline direct oral anticoagulant levels in atrial fibrillation: the MAS study. Blood Adv. 2024 Apr 23;8(8):1846-1856. doi: 10.1182/bloodadvances.2023012408. PMID 38394387

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03803579/Prot_SAP_000.pdf